CLINICAL TRIAL: NCT00553488
Title: A Mono Center Open Labeled, Randomized Study Examining the Effects of Intra-Dermal vs Subcutaneous Application of Regular Insulin or Rapid Acting Insulin Analogue on Postprandial Glycemic Excursions in Patients With Type 1 Diabetes
Brief Title: Feasibility Study of the Effect of Intra-Dermal Insulin Injection on Blood Glucose Levels After Eating
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Becton, Dickinson and Company (Industry)
Responsible Party: Laurence Hirsch, Vice-President, Global Medical Affairs, Diabetes Care, BD
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: BDT-ADD-07-002; EudraCT number 2007-003924-39
Record Dates: First submitted 2007-10-12; First posted 2007-11-05 (Estimated); Last update posted 2008-08-22 (Estimated); Status verified 2008-08

CONDITIONS: Diabetes Mellitus, Type 1
Keywords: diabetes; insulin; subcutaneous; intra-dermal; blood glucose
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus; Insulin Resistance | interventions — Insulin; Insulin, Regular, Human; Insulin Lispro

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- 1 (Active Comparator): Regular insulin SC at -17 mins
  Interventions: Drug: Regular insulin (Humulin)
- 2 (Active Comparator): Regular insulin ID at -17 mins
  Interventions: Drug: Regular insulin (Humulin)
- 3 (Active Comparator): Regular insulin ID at -2 mins
  Interventions: Drug: Regular insulin (Humulin)
- 4 (Active Comparator): Insulin lispro given SC at -2 mins
  Interventions: Drug: Insulin lispro (Humalog)
- 5 (Experimental): Insulin lispro given ID at -2 mins
  Interventions: Drug: Insulin lispro (Humalog)

INTERVENTIONS:
Drug: Regular insulin (Humulin) — Insulin will be given either subcutaneously or intra-dermally, and at two different times prior to the liquid meal (T zero). At -17 mins, regular insulin will be given either SC or ID. At -2 mins, regular insulin will be given ID; also insulin lispro will be given either SC or ID. Each patient will receive 1 injection on 5 different study days.
  Arms: 1; 2; 3
Drug: Insulin lispro (Humalog) — Insulin will be given either subcutaneously or intra-dermally, and at two different times prior to the liquid meal (T zero). At -17 mins, regular insulin will be given either SC or ID. At -2 mins, regular insulin will be given ID; also insulin lispro will be given either SC or ID. Each patient will receive 1 injection on 5 different study days.
  Arms: 4; 5

SUMMARY:
This study is to determine the effect of intra-dermal (ID) administration of regular and of rapid-acting insulin, before eating, on blood glucose levels for several hours after a standard meal (a mixed, liquid meal). Insulin will also be given normally, subcutaneously, for control or comparison purposes. The hypothesis or expectation is that ID insulin will work more quickly and control blood glucose levels better than SC injection.

DETAILED DESCRIPTION:
Previous studies have shown that intra-dermal (ID) insulin administration results in a more rapid onset of action in comparison to subcutaneous (SC) administration as measured by glucose infusion rate (GIR) under glucose clamp conditions.The aim of this study is to investigate whether ID administration of regular human insulin or rapid-acting insulin analogue leads to reduced postprandial glycemic excursions in comparison to SC application under highly standardized experimental conditions. Effects on the occurrence of hypoglycemia will also be investigated, as well as pK and pD comparisons between different insulin formulations administered ID. This is a mono-center, open-label, randomized, 5-period crossover study in patients with type 1 diabetes

ELIGIBILITY:
Inclusion Criteria:

* Type 1 diabetes for 1-15 years, on multiple daily injections (MDI) or insulin pump (CSII) in stable control with HbA1c <= 9.0%.
* Able to attend clinic for 5 different days

Exclusion Criteria:

* BMI > 32 kg/m2
* Evidence of gastroparesis or impaired renal function or lipodystrophy

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2007-09; Primary Completion 2007-12 (Actual); Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
Area Under Curve (AUC) of the blood glucose (BG) profile after the meal, with and without baseline correction. | 90 mins

SECONDARY OUTCOMES:
Maximal BG (BGmax) | Approximately 4 hours per injection
Total BG-AUC0-4 h | Approximately 4 hrs per injection
Minimal BG (BGmin, time to BGmin (tBGmin) | Approximately 4 hrs per injection
Insulin pharmacokinetics | Approximately 4 hrs per injection
Number and seriousness of adverse events | Approximately 4 hrs per injections
Vital signs, examination of insulin application | Approximately 4 hrs per injection
Time to BGmax (tBGmax) | Approximately 4 hours per injection

CONTACTS AND LOCATIONS:
Overall Officials: Christoph Kapitza, MD, Principal Investigator — Profil Institut fur Stoffwechselforschung GmbH
Locations (1):
- Profil Institut fur Stoffwechselforschung GmbH, Neuss, Germany

REFERENCES:
- [Derived] Pettis RJ, Hirsch L, Kapitza C, Nosek L, Hovelmann U, Kurth HJ, Sutter DE, Harvey NG, Heinemann L. Microneedle-based intradermal versus subcutaneous administration of regular human insulin or insulin lispro: pharmacokinetics and postprandial glycemic excursions in patients with type 1 diabetes. Diabetes Technol Ther. 2011 Apr;13(4):443-50. doi: 10.1089/dia.2010.0183. Epub 2011 Feb 28. PMID 21355716